CLINICAL TRIAL: NCT06419725
Title: Temporal Trends in Nonattendence Rate for Scheduled Outpatient Appointments.
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, LUCIA.PEREZ, Pediatrician. Non-sponsored research. Research Secretary of the University Italian Hospital of Buenos Aires., Hospital Italiano de Buenos Aires
Other Study IDs: 6922
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Patient Non Attendance to Medical Care
Keywords: No Show Patients; Patient Non Attendance; Patient absenteeism; Patient compliance
MeSH Terms: conditions — No-Show Patients; Patient Compliance

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ecological time-series study using secondary databases.

DETAILED DESCRIPTION:
A time-series study will be conducted to evaluate nonattendance over time. The unit of analysis will be the appointment.

ELIGIBILITY:
Inclusion Criteria:

* Appointments scheduled for outpatient medical care across all settings and specialties from January 1, 2016, to December 31, 2023

Exclusion Criteria:

* Cancelled appointments, including cancellations made by the patient, medical team, and the appointment management system.
* Appointments that do not correspond to scheduled in-person care (Teleconsultations,
* Appointments for walk-in demand).
* Scheduled appointments that are not for medical care (Health coverage or specialties that do not correspond to scheduled medical care, Appointments for procedures,
* Appointments for complementary exams, Appointments for treatments such as speech therapy, physiotherapy, or other therapies).
* Spontaneous overflow appointments where the patient spontaneously presents for care at that moment. These appointments cannot be absent as the present and the appointment are assigned simultaneously.
* System errors that do not correspond to actual patient medical care appointments (Duplicate cancellations, Appointments where patient and physician coincide).

Ages: 0 Years to 110 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population comprises individuals who requested at least one appointment for scheduled outpatient medical care at Hospital Italiano de Buenos Aires during the study period in any of its settings.
Sampling Method: Probability Sample
Enrollment: 13823093 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Describe the behavior over time of the nonattendance proportion in scheduled outpatient medical appointments for in-person medical care over an 8-year period (globally and by subgroups: gender, age, medical specialty, and medical coverage). | 2016 to 2023
Evaluate temporal trends and changes (joinpoints) in the absenteeism proportion in scheduled outpatient medical appointments for in-person medical care over the same period. | 2016 to 2023

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Italiano de Buenos Aires, Ciudad Autonoma de Buenos Aire, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giunta D, Briatore A, Baum A, Luna D, Waisman G, de Quiros FG. Factors associated with nonattendance at clinical medicine scheduled outpatient appointments in a university general hospital. Patient Prefer Adherence. 2013 Nov 8;7:1163-70. doi: 10.2147/PPA.S51841. eCollection 2013. PMID 24235820
- [Background] Giunta DH, Alonso Serena M, Luna D, Peroni ML, Sanchez Thomas D, Binder F, Blugerman GA, Fuentes N, Elizondo CM, Gonzalez Bernaldo de Quiros F. Association between non-attendance to outpatient clinics and emergency department consultations, hospitalizations and mortality in a Health Maintenance Organization. Int J Health Plann Manage. 2020 Sep;35(5):1140-1156. doi: 10.1002/hpm.3021. Epub 2020 Jul 9. PMID 32648278
- [Background] Carrillo GJS. Adhesión de los pacientes a las consultas de control ambulatorio. Investigación en Enfermería: Imagen y Desarrollo. 2011;9: 51-62.
- [Background] Kheirkhah P, Feng Q, Travis LM, Tavakoli-Tabasi S, Sharafkhaneh A. Prevalence, predictors and economic consequences of no-shows. BMC Health Serv Res. 2016 Jan 14;16:13. doi: 10.1186/s12913-015-1243-z. PMID 26769153
- [Background] Berg BP, Murr M, Chermak D, Woodall J, Pignone M, Sandler RS, Denton BT. Estimating the cost of no-shows and evaluating the effects of mitigation strategies. Med Decis Making. 2013 Nov;33(8):976-85. doi: 10.1177/0272989X13478194. Epub 2013 Mar 20. PMID 23515215
- [Background] Jabalera Mesa ML, Morales Asencio JM, Rivas Ruiz F, Porras Gonzalez MH. [Analysis of economic cost of missed outpatient appointments]. Rev Calid Asist. 2017 Jul-Aug;32(4):194-199. doi: 10.1016/j.cali.2017.01.004. Epub 2017 May 2. Spanish. PMID 28476506
- [Background] George A, Rubin G. Non-attendance in general practice: a systematic review and its implications for access to primary health care. Fam Pract. 2003 Apr;20(2):178-84. doi: 10.1093/fampra/20.2.178. PMID 12651793
- [Background] Wolff DL, Waldorff FB, von Plessen C, Mogensen CB, Sorensen TL, Houlind KC, Bogh SB, Rubin KH. Rate and predictors for non-attendance of patients undergoing hospital outpatient treatment for chronic diseases: a register-based cohort study. BMC Health Serv Res. 2019 Jun 14;19(1):386. doi: 10.1186/s12913-019-4208-9. PMID 31200720
- [Background] Karter AJ, Parker MM, Moffet HH, Ahmed AT, Ferrara A, Liu JY, Selby JV. Missed appointments and poor glycemic control: an opportunity to identify high-risk diabetic patients. Med Care. 2004 Feb;42(2):110-5. doi: 10.1097/01.mlr.0000109023.64650.73. PMID 14734947
- [Background] Lee RRS, Samsudin MI, Thirumoorthy T, Low LL, Kwan YH. Factors affecting follow-up non-attendance in patients with Type 2 diabetes mellitus and hypertension: a systematic review. Singapore Med J. 2019 May;60(5):216-223. doi: 10.11622/smedj.2019042. PMID 31187148
- [Background] Colubi MM, Perez-Elias MJ, Elias L, Pumares M, Muriel A, Zamora AM, Casado JL, Dronda F, Lopez D, Moreno S; SEAD Study Group. Missing scheduled visits in the outpatient clinic as a marker of short-term admissions and death. HIV Clin Trials. 2012 Sep-Oct;13(5):289-95. doi: 10.1310/hct1305-289. PMID 23134630
- [Background] Srisaenpang S, Pinitsoontorn S, Singhasivanon P, Kitayaporn D, Kaewkungwal J, Tatsanavivat P, Patjanasoontorn B, Reechaipichitkul W, Thiratakulpisan J, Srinakarin J, Srisaenpang P, Thinkamrop B, Apinyanurak C, Chindawong BO. Missed appointments at a tuberculosis clinic increased the risk of clinical treatment failure. Southeast Asian J Trop Med Public Health. 2006 Mar;37(2):345-50. PMID 17124997
- [Background] Ayten Turkcan & Lynn Nuti & Po-Ching DeLaurentis & Zhiyi Tian & Joanne Daggy & Lingsong Zhang & Mark Lawley & Laura Sands, 2013.
- [Background] Giunta DH, Alonso Serena M. Nonattendance rates of scheduled outpatient appointments in a university general hospital. Int J Health Plann Manage. 2019 Oct;34(4):1377-1385. doi: 10.1002/hpm.2797. Epub 2019 May 7. PMID 31062463
- [Background] Kim HJ, Fay MP, Feuer EJ, Midthune DN. Permutation tests for joinpoint regression with applications to cancer rates. Stat Med. 2000 Feb 15;19(3):335-51. doi: 10.1002/(sici)1097-0258(20000215)19:33.0.co;2-z. PMID 10649300
- [Background] Daniel L, Paula O, Alejandro LO, Eduardo R, Federico P, Adrián G, et al. Implementación de una Historia Clínica Electrónica Ambulatoria: El Proyecto Itálica. 6to Simposio de Informática en Salud - 32 JAIIO 2003. 2003.
- [Background] Plazzotta F, Luna D, Gonzalez Bernaldo de Quiros F. [Health information systems: integrating clinical data in different scenarios and users]. Rev Peru Med Exp Salud Publica. 2015 Apr-Jun;32(2):343-51. Spanish. PMID 26338397
- [Background] Franco M, Giussi Bordoni MV, Otero C, Landoni MC, Benitez S, Borbolla D, Luna D. Problem Oriented Medical Record: Characterizing the Use of the Problem List at Hospital Italiano de Buenos Aires. Stud Health Technol Inform. 2015;216:877. PMID 26262179
- [Background] Luna D, Franco M, Plaza C, Otero C, Wassermann S, Gambarte ML, Giunta D, Gonzalez Bernaldo de Quiros F. Accuracy of an electronic problem list from primary care providers and specialists. Stud Health Technol Inform. 2013;192:417-21. PMID 23920588
- [Background] Plazzotta F, Otero C, Luna D, de Quiros FG. Natural language processing and inference rules as strategies for updating problem list in an electronic health record. Stud Health Technol Inform. 2013;192:1163. PMID 23920937
- [Background] Torre LA, Siegel RL, Ward EM, Jemal A. International variation in lung cancer mortality rates and trends among women. Cancer Epidemiol Biomarkers Prev. 2014 Jun;23(6):1025-36. doi: 10.1158/1055-9965.EPI-13-1220. Epub 2014 May 16. PMID 24836468
- See also: National Cancer Institute. Division of Cancer Control and Population Science. Joinpoint Trend Analysis Software. — https://surveillance.cancer.gov/joinpoint/
- See also: Medidas sanitarias por la pandemia de COVID-19 en Argentina. — https://es.wikipedia.org/wiki/Medidas_sanitarias_por_la_pandemia_de_COVID-19_en_Argentina#Del_20_al_31_de_marzo
- See also: COVID-19 pandemic in Argentina. — https://en.wikipedia.org/wiki/COVID-19_pandemic_in_Argentina